CLINICAL TRIAL: NCT03208491
Title: AZ@GAME-Eco: Economic Assessment of Serious Games for the Management of Alzheimer's Disease and Related Disorders
Acronym: AZ@GAME-Eco
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16-PRME-01
Record Dates: First submitted 2017-06-26; First posted 2017-07-05 (Actual); Last update posted 2017-07-05 (Actual); Status verified 2017-05

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- serious games (Experimental)
  Interventions: Other: serious games use
- usual care (Active Comparator)
  Interventions: Other: usual care

INTERVENTIONS:
Other: serious games use — This program has enabled several SGs to be developed that allow physical and cognitive workouts to be carried out with a therapist
  Arms: serious games
Other: usual care — usual care of patient
  Arms: usual care

SUMMARY:
The main objective of AZ@GAME ECO is to evaluate the cost-utility of the management of patients suffering from Alzheimer's disease using a serious game providing cognitive and physical straining compared to a usual management. Among the secondary objectives it is important to assess the real life feasibility in different types of care structures.

DETAILED DESCRIPTION:
With the aging of the population, Alzheimer's disease and associated disorders represent a major public health challenge. To date there is no pharmacological treatment to stop the degenerative process or behavioral disorders. This explains the importance of non-pharmacological approaches to stimulate cognition, reduce behavioral disorders or improve quality of life. Non-pharmacological therapies are the central focus of care, especially for patients accommodated on a part-time basis (Day Hospital, Respite Platform) or Full-Time nursing home (EHPAD in French). TNM also holds an important place for patients living at home, and belongs to the very general framework of informal care, which is a significant cost.

In France, the cost of taking care of patients over 75 with this type of pathology is estimated between 24.2 and 30 billion euros per year, which is more than cancer or cardiovascular disease.

At the same time, new information and communication technologies (ICTs) play an increasingly important part in our daily lives and can be a support in the field of health. In this context, ICTs are of great interest for evaluation, rehabilitation and assistance. At the level of care, the aim is to propose applications to train and / or stimulate cognitions, behavior and motivation. Serious Games (SG) are part of this framework.

Az @ GAME (Alzheimer's Disease and serious games), is the winner of the e-health project 2011-2015. This program has enabled several SGs to be developed that allow physical and cognitive workouts to be carried out with a therapist. The AZ @ GAME-ECO + study is a new and innovative step as it represents the first combined evaluation of the cost and usefulness of managing patients with Alzheimer's disease using the serious Games (SG). In AZ @ GAME-ECO + SGs are a new tool for institutions involved in patient care.

OBJECTIVES The main objective of AZ@GAME ECO is to evaluate the cost-utility of the management of patients suffering from Alzheimer's disease using a serious game providing cognitive and physical straining compared to a usual management. Among the secondary objectives it is important to assess the real life feasibility in different types of care structures.

POPULATION Male or Female ≥ 60 years of age / with a diagnosis of Alzheimer's Disease or related disorders (CIM10) condition with a Mini Mental State Examination score between 12 and 24. Patients are monitored in one of the centers participating in the study (Day Hospital, nursing home, Memory Consultation).

METHOD This multi-center study involves 18 participating centers: Dependent Elderly Care Facilities (EHPAD), Day Care Centers, and Memory Centers, with the inclusion of 144 subjects (72 subjects per group and 8 subjects per center). It will be done in open form.

After randomization, the centers belonging to the intervention group use the SG for 3 months (2 sessions per week). The control group centers will be able to use the SG at the end of the study.

Medico-economic and clinical evaluations will be performed at baseline, at the end of the intervention (M3) and 3 months after the intervention (M6). An incremental cost-utility ratio will be calculated to compare the management with SG therapeutics and the usual management from a societal perspective and with a time horizon of 6 months.

BENEFITS To gain a better understanding of the medico-economic benefits and usability of a new technology to train cognitive, physical functions while promoting motivation and social engagement in Alzheimer's disease patients in situations Usual care in Daycare, Nursing home and Memory center.

PARTNERS Montpellier University Health Center / Groupe Genious / Alzheimer Innovation Association / Institut national de recherche en informatique et en automatique (INRIA) Sophia-Antipolis - STARS team

ELIGIBILITY:
Inclusion Criteria:

* Male or Female ≥ 60 years of age;
* Subjects diagnosed with Alzheimer's Disease or related disorders associated with mild to moderately severe (CIM 10)
* a score between 12 and 24 on the Mini Mental score evaluation
* Subject treated in one of the participating centers
* To have the social welfare insurance
* Signature of the free and informed consent in the case of a patient under guardianship with signature of the guardian

Exclusion Criteria:

* history of epilepsy
* major walking or balance disorder.
* Subject without freedom by judicial or administrative decision

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2017-09-30 (Estimated); Primary Completion 2018-03-30 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
cost utility ratio | at 3 months
  Measurement of the incremental cost-utility ratio of the management of patients suffering from Alzheimer's disease

IPD SHARING:
Plan to Share IPD: No